CLINICAL TRIAL: NCT03958188
Title: Assessment of an Optimized and Standardized Computerised Tomography (CT) Reading Grid for Preoperative Planning Improvement of Small Bowel Neuroendocrine Tumours (NET).
Brief Title: PreOPerative Imaging of NeuroEndocrine Tumors
Acronym: POPINET
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: POPINET
Record Dates: First submitted 2019-05-20; First posted 2019-05-21 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Neuro-endocrine Tumors; Small Intestine Cancer
Keywords: Intestinal tumors; Computerized Tomography
MeSH Terms: conditions — Intestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients who have undergone pre-operated computerized tomography (CT) imaging for a subsequently operated Neuro-endocrine tumor (NET).
  Clinical data collected for each patients:
  * Age
  * Sex
  * Symptomatology (abdominal pain, diarrhea, carcinoid flush, digestive bleeding, weight loss, occlusive syndrome)
  * Blood Chromogranine A and urinary 5-hydroxyindoleacetic acid (5-HIAA)
  * Carcinoid valvulopathy
  Interventions: Other: Standardized computerized tomography (CT) reading grid for preoperative planning

INTERVENTIONS:
Other: Standardized computerized tomography (CT) reading grid for preoperative planning — Using the standardized reading grid, the following data will be collected:
  * Small Intestine: tumor, parietal thickening, occlusive syndrome, proximity of the tumor with the ileocecal valve.
  * Mesenteric mass: presence, size, shape, contours, calcifications, enhancement, superior mesenteric arterial invasion and number of non-invaded arterial arteries.
  * Mesentery: moniliform venous dilatations, combed appearance.
  * Duodenal invasion.
  * Lymphadenopathies (Mesenteric, Right mesocolic and Retropancreatic): presence, size, shape, enhancement
  The anonymized CT exam will be reviewed by an expert radiologist and a radiology resident from imaging department of the Hospital.

SUMMARY:
Neuro-endocrine tumours (NET) are the most frequent tumours of the small intestine. In spite of their small size, these tumours have the particularity of forming mesenteric metastasis and ganglionic secondary lesions along the superior mesenteric axis, which is in close proximity to the superior mesenteric artery (SMA).

Surgery is the only curative treatment. The complete resection being a factor for good patient prognosis, risks of subsequent local complications (occlusion, bleeding) must be discussed. The limiting factor for resectability is arterial vascular invasion considering the risk of postoperative small bowel syndrome.

At the moment, the choice of imaging examination and its protocol is not standardized, nor the description of the tumoral mesenteric and ganglionic extension, especially the criteria defining a lymph node as lymphadenopathy. In addition, the complexity of SMA's anatomy and the absence of criteria for arterial invasion defining arterial invasion may lead to a misinterpretation of the preoperative imaging , and thus to an incomplete planning of the surgical procedure.

To correct this absence of radiological standardization, the investigating team has developed a reading grid for Computed Tomography (CT) aimed to facilitate preoperative planning of small bowel NET.

The main objective of the current study is to improve the semiotic description of the mesenteric and ganglionic tumoral extension of small intestine NET using a technically optimized imaging examination and a standardized reading grid in order to plan the best surgical procedure which would allow maintaining a minimal length of small intestine needed to yield a satisfying quality of life and nutritional status.

The secondary objective of this study is to evaluate the reproducibility of the standardized scanner's reading grid.

ELIGIBILITY:
Inclusion Criteria:

* Patients with small intestine neuro-endocrine tumors (NET) operated in the digestive surgical service of the University Edouard Herriot hospital of Lyon (Pr. Gilles Poncet) between the 1st of January 2014 and the 31st of March 2019,
* Having done a preoperative thoraco-abdomino-pelvic scanner with arterial and portal sequences.
* Scanner imaging, operative report and anatomo-pathological report available

Exclusion Criteria:

* no Computerized Tomography (CT) images available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients at least 18 years old with small intestine neuro-endocrine tumors (NET)
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardization of a reading grid for PreOPerative Imaging of NeuroEndocrine Tumors | 7 months
  Improve the semiological description of the mesenteric and ganglionic tumoral extension of small intestine NET using a technically optimized imaging technique with a standardized reading grid in order to plan the best surgical procedure which allows maintaining a minimal length of small intestine needed to a satisfying quality of life and nutritional status.

CONTACTS AND LOCATIONS:
Overall Officials: Romain L'Huillier, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot, Lyon, France